CLINICAL TRIAL: NCT06104046
Title: Prevalence of Seroconversion of Hepatitis c Virus Among Children With Chronic Kidney Disease on Regular Hemodialysis
Brief Title: Prevalence of Seroconversion of Hepatitis c Virus Among Children With CKD on Regular Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Zeawela, 71515,Assiut, Assiut University
Other Study IDs: seroconversion of hepatitis c
Record Dates: First submitted 2023-10-21; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
observational cross sectional study for children with chronic kidney disease who on regular hemodialysis in assiut univeristy children hospital at dialysis unit, observe prevalence of serological seroconversion of hepatitis c virus and associated risk factors

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a blood-borne pathogen that appears to be endemic in many parts of the world,the highest prevalence of HCV has been found in Egypt (17-26%) The prevalence of HCV infection is higher in most subgroups of chronic kidney disease (CKD) patients than in the general population.

As there is very little known about HCV infection in infants and children with CKD and this very limited information implies that the current guidelines do not apply directly and completely to this specific population, and as the Kidney Disease Improving Global Outcomes (KDIGO) has recommended that pediatric nephrologists and other physicians - in charge of caring for children with CKD - should carefully evaluate the extent to which the current guidelines may be extrapolated to children.

Hepatitis C virus (HCV) infection is a significant cause of morbidity and mortality in hemodialysis patients and observed as a major public health problem infecting 170 million people globally and hepatitis C virus (HCV) infection is one of the most common blood-borne infections in Egypt, a large number of egyptians are exposed to infection due to low hygiene and sterilization measures in our community The Patients who undergo maintenance hemodialysis (HD) treatment are at increased hazard of getting these infections and have a greater prevalence of HCV than the general population due to underlying impaired cellular immunity which increases their susceptibility to HCV infection the hemodialysis patients are exposed to prolonged vascular access and exposure to contaminated equipment and handling by medical staff, In addition the CKD patients require frequent blood transfusion to recover the anemia related with chronic kidney disease and this blood transfusion make a source for HCV infection The inadequate sterilization of medical equipments, invasive dialysis procedures, mode of dialysis, contaminated blood and blood products, duration of end stage kidney disease, sharing of dialysis equipment, insertion of an intravascular catheter and contact with contaminated HD equipments and supplies during hemodialysis, all these risk factors help in HCV infection in hemodialysis patients.

In this study, the prevalence of seroconversion of hepatitis c virus among children with CKD on regular hemodialysis is to be assessed and its possible risk factors related to it

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 1 year to 18 years
2. CKD children on regular hemodialysis for more than one month duration

Exclusion Criteria:

* 1-Age: less than 1 year and more than 18 years 2- CKD children who are not on regular hemodialysis and for less than one month duration

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients on regular Hemodialysis for more than one month duration in Children AUH Dialysis Unit are enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-26 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Seroconversion of Hepatitis c Virus Among Children With CKD on Regular Hemodialysis | Baseline
  determine prevalence and risk factors associated with seroconversion of hepatitis c in CKD children on regular hemodialysis

REFERENCES:
- [Background] El-Shabrawi MH, Kamal NM. Burden of pediatric hepatitis C. World J Gastroenterol. 2013 Nov 28;19(44):7880-8. doi: 10.3748/wjg.v19.i44.7880. PMID 24307782
- [Background] Kosaraju K, Faujdar SS, Singh A, Prabhu R. Hepatitis viruses in heamodialysis patients: an added insult to injury? Hepat Res Treat. 2013;2013:860514. doi: 10.1155/2013/860514. Epub 2013 Mar 6. PMID 23533739